CLINICAL TRIAL: NCT01667406
Title: The Use of the Hormone Kisspeptin in 'in Vitro Fertilisation' (IVF) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13HH0199; 2012-000154-61 (EudraCT Number)
Record Dates: First submitted 2012-08-08; First posted 2012-08-17 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Infertility
Keywords: kisspeptin; infertility; in vitro fertilisation
MeSH Terms: conditions — Infertility | interventions — Kisspeptins; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Different dose for each volunteer
Who Masked: Participant, Care Provider
Masking Description: participants and IVF physicians were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Kisspeptin-54, 1.6 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 1.6 nmol/kg
  Interventions: Drug: Kisspeptin 1.6nmol/kg
- Kisspeptin-54, 3.2 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 3.2 nmol/kg
  Interventions: Drug: Kisspeptin 3.2nmol/kg
- Kisspeptin-54, 6.4 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 6.4 nmol/kg
  Interventions: Drug: Kisspeptin 6.4nmol/kg
- Kisspeptin-54, 12.8 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 12.8 nmol/kg
  Interventions: Drug: Kisspeptin 12.8nmol/kg
- Kisspeptin-54 OHSS, 3.2 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 3.2 nmol/kg
  Interventions: Drug: Kisspeptin 3.2nmol/kg
- Kisspeptin-54 OHSS, 6.4 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 6.4 nmol/kg
  Interventions: Drug: Kisspeptin 6.4nmol/kg
- Kisspeptin-54 OHSS, 9.6 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 9.6 nmol/kg
  Interventions: Drug: Kisspeptin 9.6nmol/kg
- Kisspeptin-54 OHSS, 12.8 single (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 12.8 nmol/kg
  Interventions: Drug: Kisspeptin 12.8nmol/kg
- Kisspeptin-54 OHSS, 9.6 + 9.6 (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a trigger injection of Kisspeptin, dose of 9.6 nmol/kg and a further injection of Kisspeptin, dose of 9.6 nmol/kg 10 hours later
  Interventions: Drug: Kisspeptin 9.6 nmol/kg double
- Kisspeptin-54 OHSS, 9.6 + saline (Experimental): Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a trigger injection of Kisspeptin, dose of 9.6 nmol/kg and a further injection of saline10 hours later
  Interventions: Drug: Kisspeptin 9.6 nmol/kg + saline

INTERVENTIONS:
Drug: Kisspeptin 1.6nmol/kg — single kisspeptin dose 1.6 nmol/kg subcutaneously
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54, 1.6 single
Drug: Kisspeptin 3.2nmol/kg — single kisspeptin dose 3.2 nmol/kg subcutaneously
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54 OHSS, 3.2 single; Kisspeptin-54, 3.2 single
Drug: Kisspeptin 6.4nmol/kg — single kisspeptin dose 6.4 nmol/kg subcutaneously
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54 OHSS, 6.4 single; Kisspeptin-54, 6.4 single
Drug: Kisspeptin 9.6nmol/kg — single kisspeptin dose 9.6 nmol/kg subcutaneously
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54 OHSS, 9.6 single
Drug: Kisspeptin 12.8nmol/kg — single kisspeptin dose 12.8 nmol/kg subcutaneously
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54 OHSS, 12.8 single; Kisspeptin-54, 12.8 single
Drug: Kisspeptin 9.6 nmol/kg double — kisspeptin dose 9.6 nmol/kg given twice 10hrs apart subcutaneously
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54 OHSS, 9.6 + 9.6
Drug: Kisspeptin 9.6 nmol/kg + saline — kisspeptin dose 9.6 nmol/kg subcutaneously and saline subcutaneously, 10hrs apart
  Other Names: kisspeptin-54
  Arms: Kisspeptin-54 OHSS, 9.6 + saline

SUMMARY:
We want to find out if kisspeptin is successful in stimulating oocyte maturation when it is used as a 'trigger' injection during IVF therapy for infertility.

DETAILED DESCRIPTION:
Participants in the study will have a standard Gonadotrophin Releasing Hormone (GnRH) antagonist IVF cycle, but instead of having a trigger injection of hCG (human chorionic gonadotrophin) they will be randomised to receive one of 4 doses of kisspeptin injection.

Oocytes will be retrieved and graded by an embryologist to see whether or not they have matured.

The reproductive hormones Luteinising hormone, follicle stimulating hormone, oestradiol and progesterone will also be measured

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 34 years
* Body mass index between 18 and 29 kg/m2
* Stable body weight for at least 3 months
* Normal early menstrual cycle follicular phase serum FSH concentration
* Serum anti-Mullerian hormone (AMH) > 40pmol/L
* No more than one previous IVF treatment cycle
* Both ovaries intact

Exclusion Criteria:

History of any medical, psychological or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or potentially cause harm to the volunteer

* Without access at home to a telephone, or other factor likely to interfere with ability to participate reliably in the study
* Treatment with an investigational drug within the preceding 2 months
* Donated blood during the preceding 3 months or intention to do so before the end of the study
* Previous poor response to IVF treatment

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — woman undergoing IVF treatment
Enrollment: 175 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waljit S Dhillo, PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be presented in anonymised groups

REFERENCES:
- [Result] Jayasena CN, Abbara A, Comninos AN, Nijher GM, Christopoulos G, Narayanaswamy S, Izzi-Engbeaya C, Sridharan M, Mason AJ, Warwick J, Ashby D, Ghatei MA, Bloom SR, Carby A, Trew GH, Dhillo WS. Kisspeptin-54 triggers egg maturation in women undergoing in vitro fertilization. J Clin Invest. 2014 Aug;124(8):3667-77. doi: 10.1172/JCI75730. Epub 2014 Jul 18. PMID 25036713
- [Result] Abbara A, Clarke S, Islam R, Prague JK, Comninos AN, Narayanaswamy S, Papadopoulou D, Roberts R, Izzi-Engbeaya C, Ratnasabapathy R, Nesbitt A, Vimalesvaran S, Salim R, Lavery SA, Bloom SR, Huson L, Trew GH, Dhillo WS. A second dose of kisspeptin-54 improves oocyte maturation in women at high risk of ovarian hyperstimulation syndrome: a Phase 2 randomized controlled trial. Hum Reprod. 2017 Sep 1;32(9):1915-1924. doi: 10.1093/humrep/dex253. PMID 28854728
- [Result] Abbara A, Jayasena CN, Christopoulos G, Narayanaswamy S, Izzi-Engbeaya C, Nijher GM, Comninos AN, Peters D, Buckley A, Ratnasabapathy R, Prague JK, Salim R, Lavery SA, Bloom SR, Szigeti M, Ashby DA, Trew GH, Dhillo WS. Efficacy of Kisspeptin-54 to Trigger Oocyte Maturation in Women at High Risk of Ovarian Hyperstimulation Syndrome (OHSS) During In Vitro Fertilization (IVF) Therapy. J Clin Endocrinol Metab. 2015 Sep;100(9):3322-31. doi: 10.1210/jc.2015-2332. Epub 2015 Jul 20. PMID 26192876
- [Derived] Abbara A, Islam R, Clarke SA, Jeffers L, Christopoulos G, Comninos AN, Salim R, Lavery SA, Vuong TNL, Humaidan P, Kelsey TW, Trew GH, Dhillo WS. Clinical parameters of ovarian hyperstimulation syndrome following different hormonal triggers of oocyte maturation in IVF treatment. Clin Endocrinol (Oxf). 2018 Jun;88(6):920-927. doi: 10.1111/cen.13569. Epub 2018 Mar 6. PMID 29446481
- [Derived] Owens LA, Abbara A, Lerner A, O'floinn S, Christopoulos G, Khanjani S, Islam R, Hardy K, Hanyaloglu AC, Lavery SA, Dhillo WS, Franks S. The direct and indirect effects of kisspeptin-54 on granulosa lutein cell function. Hum Reprod. 2018 Feb 1;33(2):292-302. doi: 10.1093/humrep/dex357. PMID 29206944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parallel study, volunteers received only one type of dose
Groups:
- Kisspeptin-54 1.6 Single: Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 1.6 nmol/kg
- Kispeptin-54 3.2 Single: Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 3.2 nmol/kg
- Kisspeptin-54 6.4 Single: Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 6.4 nmol/kg
- Kisspeptin-54 12.8 Single: Participant undergoing in vitro fertilisation (IVF) treatment will receive a single trigger injection of Kisspeptin, dose of 12.8 nmol/kg
- OHSS - Kisspeptin-54 3.2 Single: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 3.2 nmol/kg
- OHSS - Kisspeptin-54 6.4 Single: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 6.4 nmol/kg
- OHSS - Kisspeptin-54 9.6 Single: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 9.6 nmol/kg
- OHSS - Kisspeptin-54 12.8 Single: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a single trigger injection of Kisspeptin, dose of 12.8 nmol/kg
- Kisspeptin-54 9.6 + 9.6: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a trigger injection of Kisspeptin, dose of 9.6 nmol/kg and a further injection of Kisspeptin, dose of 9.6 nmol/kg 10 hours later
- Kisspeptin-54 9.6 + Saline: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a trigger injection of Kisspeptin, dose of 9.6 nmol/kg and a further injection of saline10 hours later
Period: Overall Study
Arm/Group | Kisspeptin-54 1.6 Single | Kispeptin-54 3.2 Single | Kisspeptin-54 6.4 Single | Kisspeptin-54 12.8 Single | OHSS - Kisspeptin-54 3.2 Single | OHSS - Kisspeptin-54 6.4 Single | OHSS - Kisspeptin-54 9.6 Single | OHSS - Kisspeptin-54 12.8 Single | Kisspeptin-54 9.6 + 9.6 | Kisspeptin-54 9.6 + Saline
Started | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
Completed | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kisspeptin-54 1.6 Single | Kispeptin-54 3.2 Single | Kisspeptin-54 6.4 Single | Kisspeptin-54 12.8 Single | OHSS - Kisspeptin-54 3.2 Single | OHSS - Kisspeptin-54 6.4 Single | OHSS - Kisspeptin-54 9.6 Single | OHSS - Kisspeptin-54 12.8 Single | Kisspeptin-54 9.6 + 9.6 | Kisspeptin-54 9.6 + Saline | Total
Number analyzed (Participants) | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31 | 175
Age, Customized [Median (Inter-Quartile Range); unit: years] | 30 [28 to 32] | 31 [31 to 32] | 32 [29 to 34] | 30 [29 to 33] | 30 [28 to 31] | 30 [28 to 31] | 32 [30 to 33] | 31 [28 to 34] | 30.9 [29.1 to 32.6] | 31.2 [27.9 to 33.4] | 31.1 [29 to 32.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31 | 175
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31 | 175
BMI 18-29 [Mean (Standard Deviation); unit: kg/m^2] | 23 (0.74) | 22 (0.74) | 22 (2.22) | 23 (1.48) | 22 (2.96) | 22 (5.19) | 25 (2.96) | 24 (5.19) | 26.6 (4.52) | 23.9 (4.074) | 23.35 (1.547)
Anti-mullerian hormone (AMH) [Median (Standard Deviation); unit: pmol/L] | 21 (3.70) | 13 (5.19) | 18 (8.89) | 21 (9.63) | 35 (15.56) | 48 (22.22) | 66 (20.0) | 53 (18.52) | 44 (16.15) | 52.4 (33.33) | 37.12 (18.11)
Antral Follicle Count (AFC) [Median (Standard Deviation); unit: Follicles] | 30 (2.22) | 24 (5.93) | 20 (7.41) | 20 (6.67) | 35 (15.56) | 48 (2.22) | 66 (20) | 53 (18.52) | 33 (8.89) | 39 (16.30) | 36.8 (15.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Oocyte Maturation
Description: This was assessed by oocyte yield (percentage of mature [metaphase 2; M2] oocytes collected from the number of follicles ≥ 14 mm on final ultrasound scan prior to kisspeptin-54 trigger administration
Time Frame: 36 hours post Kisspeptin-54 trigger injection
Measure: Mean (Standard Deviation); unit: percentage of expected oocyte yield
Groups:
- Kisspeptin-54 1.6 Nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 1.6nmol/kg as a trigger injection.
- Kisspeptin-54 3.2nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 3.2nmol/kg as a trigger injection.
- Kisspeptin-54 6.4 Nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 6.4nmol/kg as a trigger injection.
- Kisspeptin-54 12.8nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 12.8nmol/kg as a trigger injection.
- Kisspeptin-54, OHSS 3.2nmol/Kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 3.2nmol/kg as a trigger injection.
- Kisspeptin-54, OHSS 6.4nmol/Kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 6.4nmol/kg as a trigger injection.
- Kisspeptin-54, OHSS 9.6nmol/Kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 9.6nmol/kg as a trigger injection.
- Kisspeptin-54, OHSS 12.8nmol/Kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 12.8nmol/kg as a trigger injection.
Arm/Group | Kisspeptin-54 1.6 Nmol/kg Single | Kisspeptin-54 3.2nmol/kg Single | Kisspeptin-54 6.4 Nmol/kg Single | Kisspeptin-54 12.8nmol/kg Single | Kisspeptin-54, OHSS 3.2nmol/Kg Single | Kisspeptin-54, OHSS 6.4nmol/Kg Single | Kisspeptin-54, OHSS 9.6nmol/Kg Single | Kisspeptin-54, OHSS 12.8nmol/Kg Single | Kisspeptin-54 OHSS, 9.6 + 9.6 | Kisspeptin-54 OHSS, 9.6 + Saline
Number analyzed (Participants) | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
percentage of expected oocyte yield | 49 (29) | 36 (18) | 76 (49) | 103 (53) | 53 (41) | 86 (49) | 86 (74) | 121 (119) | 55 (18) | 46 (22)
Statistical Analysis 1: Comparison: Kisspeptin-54 1.6 Nmol/kg Single vs Kisspeptin-54 3.2nmol/kg Single vs Kisspeptin-54 6.4 Nmol/kg Single vs Kisspeptin-54 12.8nmol/kg Single; Data presented using descriptive statistics. Confidence intervals were derived for the difference between the means of different doses; Test type: Other — Fishers exact conditional test was used to confirm significance; Mean Difference (Final Values) = 6
Statistical Analysis 2: Comparison: Kisspeptin-54, OHSS 3.2nmol/Kg Single vs Kisspeptin-54, OHSS 6.4nmol/Kg Single vs Kisspeptin-54, OHSS 9.6nmol/Kg Single; Phase 2; Test type: Other; p < 0.05, Fisher Exact
Statistical Analysis 3: Comparison: Kisspeptin-54 OHSS, 9.6 + 9.6 vs Kisspeptin-54 OHSS, 9.6 + Saline; Phase 3; Test type: Other; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.05 — Estimate of difference in success rates and estimate of odds ratio for success were derived, with P value comparing 2 treatment groups, 95% conﬁdence intervals

2. Secondary Outcome: Biochemical Pregnancy
Description: Number of participants achieving biochemical pregnancy by serum βhCG > 10 mIU/mL
Time Frame: 11 days after embryo transfer
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- KP-54 1.6nmol/kg Single: Participants undergoing IV treatment with trigger dose 1.6nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 3.2nmol/kg Single: Participants undergoing IV treatment with trigger dose 3.2nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 6.4nmol/kg Single: Participants undergoing IV treatment with trigger dose 6.4nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 12.8nmol/kg Single: Participants undergoing IV treatment with trigger dose 12.8nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 OHSS 3.2nmol/kg Single: Participants, at high risk of ovarian hyper-stimulation syndrome, undergoing IV treatment with trigger dose 3.2nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 OHSS 6.4nmol/kg Single: Participants, at high risk of ovarian hyper-stimulation syndrome, undergoing IV treatment with trigger dose 6.4nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 OHSS 9.6nmol/kg: Participants, at high risk of ovarian hyper-stimulation syndrome, undergoing IV treatment with trigger dose 9.6nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 OHSS 12.8nmol/kg Single: Participants, at high risk of ovarian hyper-stimulation syndrome, undergoing IV treatment with trigger dose 12.8nmol/kg had blood level of luteinising hormone (LH) measured at T=0
- KP-54 OHSS 9.6 +9.6 Nmol/kg: Participants, at high risk of ovarian hyper-stimulation syndrome, undergoing IV treatment with trigger dose 9.6nmol/kg followed by another injection of KP-54 9.6nmol/kg 10 hours later, had blood level of luteinising hormone (LH) measured at T=0
- KP-54 OHSS 9.6 + Saline: Participants, at high risk of ovarian hyper-stimulation syndrome, undergoing IV treatment with trigger dose 9.6nmol/kg followed by another injection of saline10 hours later, had blood level of luteinising hormone (LH) measured at T=0
Arm/Group | KP-54 1.6nmol/kg Single | KP-54 3.2nmol/kg Single | KP-54 6.4nmol/kg Single | KP-54 12.8nmol/kg Single | KP-54 OHSS 3.2nmol/kg Single | KP-54 OHSS 6.4nmol/kg Single | KP-54 OHSS 9.6nmol/kg | KP-54 OHSS 12.8nmol/kg Single | KP-54 OHSS 9.6 +9.6 Nmol/kg | KP-54 OHSS 9.6 + Saline
Number analyzed (Participants) | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
Participants | 1 | 1 | 11 | 8 | 1 | 10 | 10 | 6 | 16 | 10
Statistical Analysis 1: Comparison: KP-54 1.6nmol/kg Single vs KP-54 3.2nmol/kg Single vs KP-54 6.4nmol/kg Single vs KP-54 12.8nmol/kg Single vs KP-54 OHSS 3.2nmol/kg Single vs KP-54 OHSS 6.4nmol/kg Single vs KP-54 OHSS 9.6nmol/kg vs KP-54 OHSS 12.8nmol/kg Single vs KP-54 OHSS 9.6 +9.6 Nmol/kg vs KP-54 OHSS 9.6 + Saline; Study data were summarised using standard descriptive methods. Continuous variables following a normal distribution have been summarised using mean and SD; Test type: Other — secondary outcomes were analysed using descriptive statistics; secondary outcomes were analysed using descriptive statistics

3. Secondary Outcome: Occurrence of OHSS
Description: Women were routinely screened for the development of early OHSS and late OHSS. Women were screened by symptoms, blood analysis, and ultrasound parameters
Time Frame: 11 days following embryo transfer
Population: Occurence of OHSS was not analysed in the groups where number of participants analysed is zero as this first phase was to test only the hypothesis that kisspeptin-54 could be used to trigger egg maturation in women undergoing in vitro fertilization therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Kisspeptin-54, 1.6 Single | Kisspeptin-54, 3.2 Single | Kisspeptin-54, 6.4 Single | Kisspeptin-54, 12.8 Single | Kisspeptin-54 OHSS, 3.2 Single | Kisspeptin-54 OHSS, 6.4 Single | Kisspeptin-54 OHSS, 9.6 Single | Kisspeptin-54 OHSS, 12.8 Single | Kisspeptin-54 OHSS, 9.6 + 9.6 | Kisspeptin-54 OHSS, 9.6 + Saline
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 20 | 15 | 20 | 31 | 31
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1

4. Secondary Outcome: Fertilization Rate
Description: Percentage of M2 oocytes that fertilize to form two pronuclear [2PN] zygotes following intracytoplasmic injection with sperm [ICSI]
Time Frame: 3 days after oocyte retrieval
Population: All participants
Measure: Mean (Standard Deviation); unit: percentage of 2PN zygotes
Arm/Group | Kisspeptin-54 1.6 Single | Kispeptin-54 3.2 Single | Kisspeptin-54 6.4 Single | Kisspeptin-54 12.8 Single | OHSS - Kisspeptin-54 3.2 Single | OHSS - Kisspeptin-54 6.4 Single | OHSS - Kisspeptin-54 9.6 Single | OHSS - Kisspeptin-54 12.8 Single | Kisspeptin-54 9.6 + 9.6 | Kisspeptin-54 9.6 + Saline
Number analyzed (Participants) | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
percentage of 2PN zygotes | 14.28 (20.20) | 58.33 (30.04) | 66.94 (26.98) | 76.01 (26.28) | 68 (39) | 76 (29) | 74 (33) | 73 (21) | 78.6 (26.2) | 78.9 (37.7)

5. Secondary Outcome: Embryo Formation
Description: All embryos were graded at day 3 by an independent embryologist, blinded to doses of kisspeptin administered, using the British Fertility Society and Association of Clinical Embryologist embryo grading scheme for cleavage stage embryos, which describes embryos based on cell number, blastomere size, and fragmentation
Time Frame: 3 days after oocyte retrieval
Population: All participants
Measure: Mean (Standard Deviation); unit: formed embryos
Arm/Group | Kisspeptin-54 1.6 Single | Kispeptin-54 3.2 Single | Kisspeptin-54 6.4 Single | Kisspeptin-54 12.8 Single | OHSS - Kisspeptin-54 3.2 Single | OHSS - Kisspeptin-54 6.4 Single | OHSS - Kisspeptin-54 9.6 Single | OHSS - Kisspeptin-54 12.8 Single | Kisspeptin-54 9.6 + 9.6 | Kisspeptin-54 9.6 + Saline
Number analyzed (Participants) | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
formed embryos | 0 (0) | 2.33 (2.31) | 3.8 (2.7) | 4.5 (2.7) | 5.8 (4.8) | 9.4 (7) | 6.5 (5.6) | 11.1 (8.4) | 6 (4.44) | 5 (3.70)

6. Secondary Outcome: Number of Participants With Clinical Pregnancy
Description: Intrauterine gestational sac with heartbeat on ultrasound at 6 weeks' gestation
Time Frame: 6 weeks after embryo transfer
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Kisspeptin-54 1.6 Single | Kispeptin-54 3.2 Single | Kisspeptin-54 6.4 Single | Kisspeptin-54 12.8 Single | OHSS - Kisspeptin-54 3.2 Single | OHSS - Kisspeptin-54 6.4 Single | OHSS - Kisspeptin-54 9.6 Single | OHSS - Kisspeptin-54 12.8 Single | Kisspeptin-54 9.6 + 9.6 | Kisspeptin-54 9.6 + Saline
Number analyzed (Participants) | 2 | 3 | 24 | 24 | 5 | 20 | 15 | 20 | 31 | 31
Participants | 1 | 0 | 7 | 4 | 1 | 10 | 10 | 6 | 7 | 12

ADVERSE EVENTS:
Time Frame: 4 years
Groups:
- KP-54 1.6nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 1.6nmol/kg as a trigger injection.
- KP-54 3.2nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 3.2nmol/kg as a trigger injection.
- KP-54 6.4nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 6.4nmol/kg as a trigger injection.
- KP-54 12.8nmol/kg Single: Participants undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 12.8nmol/kg as a trigger injection.
- KP-54 OHSS 3.2nmol/kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 3.2nmol/kg as a trigger injection.
- KP-54 OHSS 6.4nmol/kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 6.4nmol/kg as a trigger injection.
- KP-54 OHSS 9.6nmol/kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 9.6nmol/kg as a trigger injection.
- KP-54 OHSS 12.8nmol/kg Single: Participants with a high risk of ovarian hyper-stimulation syndrome (OHSS), undergoing IVF treatment received a single injection of Kisspeptin-54, at a dose of 12.8nmol/kg as a trigger injection.
- KP-54 OHSS 9.6 + 9.6 Nmol/kg: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a trigger injection of Kisspeptin, dose of 9.6 nmol/kg and a further injection of Kisspeptin, dose of 9.6 nmol/kg 10 hours later
- KP-54 OHSS 9.6nmol/kg + Saline: Participant undergoing in vitro fertilisation (IVF) treatment and who is at high risk of ovarian hyper stimulation syndrome (OHSS) will receive a trigger injection of Kisspeptin, dose of 9.6 nmol/kg and a further injection of saline10 hours later
Arm/Group | KP-54 1.6nmol/kg Single | KP-54 3.2nmol/kg Single | KP-54 6.4nmol/kg Single | KP-54 12.8nmol/kg Single | KP-54 OHSS 3.2nmol/kg Single | KP-54 OHSS 6.4nmol/kg Single | KP-54 OHSS 9.6nmol/kg Single | KP-54 OHSS 12.8nmol/kg Single | KP-54 OHSS 9.6 + 9.6 Nmol/kg | KP-54 OHSS 9.6nmol/kg + Saline
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/24 | 0/24 | 0/5 | 0/20 | 0/15 | 0/20 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 1/24 | 2/24 | 0/5 | 1/20 | 2/15 | 2/20 | 0/31 | 1/31
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/24 | 0/24 | 0/5 | 0/20 | 0/15 | 0/20 | 0/31 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KP-54 1.6nmol/kg Single (N=2) | KP-54 3.2nmol/kg Single (N=3) | KP-54 6.4nmol/kg Single (N=24) | KP-54 12.8nmol/kg Single (N=24) | KP-54 OHSS 3.2nmol/kg Single (N=5) | KP-54 OHSS 6.4nmol/kg Single (N=20) | KP-54 OHSS 9.6nmol/kg Single (N=15) | KP-54 OHSS 12.8nmol/kg Single (N=20) | KP-54 OHSS 9.6 + 9.6 Nmol/kg (N=31) | KP-54 OHSS 9.6nmol/kg + Saline (N=31)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Heterotopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Still birth (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-02-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT01667406/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT01667406/SAP_001.pdf